CLINICAL TRIAL: NCT00282295
Title: Safety & Immunogenicity of a Booster Dose of dTPa Vaccine (Boostrix®) Co-admnd. With Aventis Pasteur's Meningococcal (Serogroups A, C, Y and W-135) Polysaccharide Vaccine (Menactra™) vs Admn. of Either Vaccine Alone in Healthy Adolescents
Brief Title: US-licensed Combined Vaccine Against Tetanus & Diphtheria, Given With US-licensed Vaccine Against Meningococcal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 105753
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-06

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria
Keywords: tetanus; pertussis; Prophylaxis; meningococcus; diptheria
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Boostrix; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Boostrix + Menactra Group (Experimental): Subjects, 11 through 18 years of age, received a booster dose of Boostrix® co-administered with Menactra™ at Day 0. The Boostrix® vaccine was administered intramuscularly into the left deltoid region and Menactra™ vaccine was administered intramuscularly into the right deltoid region.
  Interventions: Biological: Boostrix®; Biological: Menactra™
- Boostrix-Menactra Group (Experimental): Subjects, 11 through 18 years of age, received one dose of Boostrix® vaccine at Day 0, followed by one dose of Menactra™ vaccine at Month 1. Both vaccines were administered intramuscularly into the left deltoid region.
  Interventions: Biological: Boostrix®; Biological: Menactra™
- Menactra-Boostrix Group (Experimental): Subjects, 11 through 18 years of age, received one dose of Menactra™ vaccine at Day 0 followed by one dose of Boostrix® vaccine at Month 1. Both vaccines were administered intramuscularly into the left deltoid region.
  Interventions: Biological: Boostrix®; Biological: Menactra™

INTERVENTIONS:
Biological: Boostrix® — GlaxoSmithKline (GSK) Biologicals' registered tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed, containing 0.3 mg aluminum.
Biological: Menactra™ — Aventis Pasteur's me ningococcal polysaccharide diphtheria toxoid conjugate vaccine containing Neisseria meningitidis serogroups, A, C, Y and W-135.

SUMMARY:
New immunization recommendations in the US include vaccination of adolescents against pertussis and meningococcal disease. The Advisory Committee on Immunization Practices of the Centers for Disease Control and Prevention recommends that Tdap (Tetanus Toxoid, Reduced Diphtheria Toxoid And Acellular Pertussis Vaccine Adsorbed) and MCV4 (Meningococcal conjugate vaccine against serotypes A, C, Y and W-135) vaccines be administered to adolescents at the same office visit if vaccination with both vaccines is indicated. Therefore, this study is designed to evaluate the safety and immunogenicity of a booster vaccination with Boostrix co-administered with Menactra as compared to the administration of either vaccine alone in healthy adolescents 11 - 18 years of age.

DETAILED DESCRIPTION:
A phase IV, randomized, partially blinded multicenter study to evaluate the safety and immunogenicity of a booster vaccination with GlaxoSmithKline's tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine, adsorbed [Tdap Boostrix®] co-administered intramuscularly with Aventis-Pasteur's meningococcal (serogroups A, C, Y and W-135) polysaccharide diphtheria toxoid conjugate vaccine (Menactra™) as compared to the administration of either vaccine alone in healthy adolescents 11-18 years of age. "Experimental design: Prospective, randomized, controlled multicenter study with three groups:

Group 1: Boostrix + Menactra on Day 0, blood samples at Month 0 and Month 1 Group 2: Boostrix on Day 0, Menactra at Month 1, blood samples at Month 0, Month 1, and Month 2 Group 3: Menactra on Day 0, Boostrix at Month 1, blood samples at Month 0, Month 1 and Month 2 Treatment allocation: randomized 1:1:1 Type of study: self-contained Duration of the study: Approximately one month for each subject in Group 1 and approximately two months for each subject in the Group 2 and Group 3."

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as established by medical history and history-directed physical examination before entering into the study.
* Previously completed routine childhood vaccinations against diphtheria, tetanus and pertussis diseases according to the recommended vaccination schedule at the time.
* Females of childbearing potential at the time of study entry are required to have a negative pregnancy test prior to administration of the dose of vaccine and are required to be abstinent or use adequate contraceptive precautions for one month prior to vaccination. Subjects also are required to agree to continue such precautions for two months after vaccination.

Exclusion Criteria:

* Administration of a pre-school booster of DTP vaccine within the previous 5 years
* Administration of a diphteria-tetanus (Td) booster within the previous 5 years
* Previous vaccination against N. meningitidis
* Hypersensitivity to latex
* History of serious allergic reaction (e.g. anaphylaxis) following any other tetanus toxoid, diphteria toxoid or pertussis-containing vaccine or any component of the study vaccines
* History of encephalopathy (e.g. coma, decreased level of consciousness, prolonged seizures) within seven days of administration of a previous dose of pertussis vaccine taht is not attributable to another identifiable cause
* Progressive neurologic disorder, uncontrolled epilepsy or progressive encephalopathy: pertussis vaccine should not be administered to individuals with these conditions until a treatment regimen has been established and the condition has stabilized
* Previous history of Guillain-Barré syndrome

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1344 (Actual)
Dates: Start 2006-01-25 (Actual); Primary Completion 2006-08-08 (Actual); Study Completion 2006-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Pittsford, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, University Heights, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Friedland et al. Immunogenicity of coadministered Tdap and MCV4 vaccines compared to separately administered vaccines. Accepted for poster presentation at ICAAC 2007
- [Result] Weston et al. Reactogenicity of concomitant and separately administered Tdap and MCV4 vaccines. Accepted for poster presentation at ICAAC 2007
- [Derived] Weston WM, Friedland LR, Wu X, Howe B. Immunogenicity and reactogenicity of co-administered tetanus-diphtheria-acellular pertussis (Tdap) and tetravalent meningococcal conjugate (MCV4) vaccines compared to their separate administration. Vaccine. 2011 Jan 29;29(5):1017-22. doi: 10.1016/j.vaccine.2010.11.057. Epub 2010 Dec 4. PMID 21134450
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 105753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 1344 subjects enrolled, only 1341 were vaccinated.
Period: Overall Study
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Started | 446 | 446 | 449
Completed | 443 | 429 | 441
Not Completed | 3 | 17 | 8
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Serious Adverse Events | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 6 | 4
Not completed — Lost to Follow-up | 1 | 7 | 2
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group | Total
Number analyzed (Participants) | 446 | 446 | 449 | 1341
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.5 (2.31) | 13.2 (2.07) | 13.4 (2.27) | 13.37 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 233 | 223 | 666
  Male | 236 | 213 | 226 | 675

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: Cut-off values assessed were greater than or equal to 1.0 international units per milliliter (IU/mL).
Time Frame: At Month 1 (post Boostrix vaccination)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects with immunogenicity data available and (&) randomization code not broken who had received at least 1 dose of study vaccine (known administration site) & had not received a vaccine not specified or forbidden by the protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Boostrix + Menactra Group: Subjects, 11 through 18 years of age, received a booster dose of Boostrix co-administered with Menactra at Day 0. The Boostrix vaccine was administered intramuscularly into the left deltoid region and Menactra vaccine was administered intramuscularly into the right deltoid region.
- Boostrix-Menactra Group: Subjects, 11 through 18 years of age, received one dose of Boostrix vaccine at Day 0, followed by one dose of Menactra vaccine at Month 1. Both vaccines were administered intramuscularly into the left deltoid region.
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group
Number analyzed (Participants) | 428 | 415
Participants
  Anti-D | 427 | 405
  Anti-T | 425 | 412
Statistical Analysis 1: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; The non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to the percentage of subjects with anti-diphtheria toxoid (anti-D) antibody concentrations equal to or greater than (≥) 1.0 IU/mL one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was greater than (>) the pre-defined limit of -10%; Difference = 2.18, 95% CI 2-sided [0.79 to 4.17]
Statistical Analysis 2: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; Non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared toBoostrix® vaccine administered alone at Month 0 with respect to the percentage of subjects with anti-tetanus toxoid (anti-T) antibody concentrations equal to or greater than (≥) 1.0 IU/mL one month after vaccination; Test type: Non-Inferiority or Equivalence — The non-inferiority objective was demonstrated if the lower limit was greater than (>) the pre-defined limit of -10%; Difference = 0.02, 95% CI 2-sided [-1.4 to 1.48]

2. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations were presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 1 (post Boostrix vaccination)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity,which included all evaluable subjects with immunogenicity data available & randomization code not broken who had received at least 1 dose of study vaccine (known administration site) & had not received a vaccine not specified or forbidden by the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group
Number analyzed (Participants) | 428 | 415
EL.U/mL
  Anti-PT: number analyzed (Participants) | 424 | 413
  Anti-PT | 63.9 [58.6 to 69.7] | 74.3 [67.9 to 81.3]
  Anti-FHA: number analyzed (Participants) | 426 | 414
  Anti-FHA | 444.8 [415.0 to 476.7] | 575.8 [532.8 to 622.1]
  Anti-PRN | 253.4 [224.8 to 285.6] | 366.0 [321.6 to 416.6]
Statistical Analysis 1: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; Non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to anti-pertussis toxoid (anti-PT) geometric mean antibody concentrations (GMCs) one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was greater than (>) the pre-defined limit of 0.67; Adjusted GMC ratio = 0.93, 95% CI 2-sided [0.84 to 1.03]
Statistical Analysis 2: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; Non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to anti-filamentous hemagglutinin (anti-FHA) GMCs one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was > the pre-defined limit of 0.67; Adjusted GMC ratio = 0.76, 95% CI 2-sided [0.69 to 0.84]
Statistical Analysis 3: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; To demonstrate the non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to anti-pertactin (anti-PRN) GMCs one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was > the pre-defined limit of 0.67; Adjusted GMC ratio = 0.63, 95% CI 2-sided [0.54 to 0.72]

3. Primary Outcome: Number of Subjects With Booster Responses for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies
Description: Booster responses for anti-PT, anti-FHA and anti-PRN antibodies were defined as:
  for initially seronegative subjects (pre-vaccination concentration below the cut-off concentration of 5 EL.U/mL): antibody concentrations at least four times the cut-off (postvaccination concentration ≥ 20 EL.U/mL) one month after vaccination with the Boostrix vaccine; for initially seropositive subjects with pre-vaccination concentration ≥5 EL.U/mL and < 20 EL.U/mL: an increase in antibody concentrations of at least four times the pre-vaccination concentration, one month after vaccination with the Boostrix vaccine; and for initially seropositive subjects with pre-vaccination concentration ≥ 20 EL.U/mL: an increase in antibody concentrations of at least two times the pre-vaccination concentration one month after vaccination with the Boostrix vaccine.
Time Frame: At Month 1 (post Boostrix vaccination)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects with immunogenicity data available & randomization code not broken who had received at least 1 dose of study vaccine (known administration site) & had not received a vaccine not specified or forbidden by the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group
Number analyzed (Participants) | 427 | 414
Participants
  Anti-PT, Total: number analyzed (Participants) | 418 | 409
  Anti-PT, Total | 322 | 333
  Anti-FHA, Total: number analyzed (Participants) | 423 | 411
  Anti-FHA, Total | 385 | 388
  Anti-PRN, Total | 398 | 394
Statistical Analysis 1: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; Non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to a booster response to PT one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was > the pre-defined limit of -10%; Difference in booster response rate = -4.38, 95% CI 2-sided [-9.91 to 1.15]
Statistical Analysis 2: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; Non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to a booster response to FHA one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was > the pre-defined limit of -10%; Difference in booster response rate = -3.39, 95% CI 2-sided [-7.03 to 0.15]
Statistical Analysis 3: Comparison: Boostrix + Menactra Group vs Boostrix-Menactra Group; To demonstrate the non-inferiority of Boostrix® vaccine co-administered with Menactra™ vaccine compared to Boostrix® vaccine administered alone at Month 0 with respect to a booster response to PRN one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was > the pre-defined limit of -10%; Difference in booster response rate = -1.96, 95% CI 2-sided [-5.25 to -1.25]

4. Primary Outcome: Number of Subjects With Vaccine Responses for Serum Bactericidal Assay Against Neisseria Meningitidis Serogroups A (rSBA-MenA), C (rSBA-MenC), Y (rSBA-MenY) and W-135 (rSBA-MenW-135)
Description: Vaccine responses for rSBA-MenA, rSBA-MenC, rSBA-MenY and rSBA-MenW-135 antibodies were defined as: for initially seronegative subjects (pre-vaccination concentration below the cut-off titer of 8): antibody titers at least four times the cut-off (post-vaccination concentration ≥ 32) one month after vaccination with Menactra vaccination; and for initially seropositive subjects (pre-vaccination titer ≥ 8): antibody titers at least four times the pre-vaccination antibody titers, one month after vaccination with Menactra vaccine.
Time Frame: One month post Boostrix vaccination ((Month 1 for Boostrix + Menactra Group and Month 2 for Menactra-Boostrix Group)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Boostrix + Menactra Group: Subjects, 11 through 18 years of age, received a booster dose of Boostrix co-admisistered with Menactra at Day 0. The Boostrix vaccine was administered intramuscularly into the left deltoid region and Menactra vaccine was administered intramuscularly into the right deltoid region.
- Menactra-Boostrix Group: Subjects, 11 through 18 years of age, received one dose of Menactra vaccine at Day 0 followed by one dose of Boostrix vaccine at Month 1. Both vaccines were administered intramuscularly into the left deltoid region.
Arm/Group | Boostrix + Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 413 | 418
Participants
  rSBA-MenA, Total: number analyzed (Participants) | 372 | 370
  rSBA-MenA, Total | 329 | 328
  rSBA-MenC, Total: number analyzed (Participants) | 413 | 413
  rSBA-MenC, Total | 390 | 383
  rSBA-MenY, Total: number analyzed (Participants) | 413 | 409
  rSBA-MenY, Total | 369 | 358
  rSBA-MenW-135, Total | 404 | 394
Statistical Analysis 1: Comparison: Boostrix + Menactra Group vs Menactra-Boostrix Group; Non-inferiority of Menactra™ vaccine co-administered with Boostrix® vaccinecompared to Menactra™ vaccine administered alone at Month 0 with respect to a vaccine responseto meningococcal serogroup A one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was greater than the pre-defined limit of -10%; Difference in vaccine response rate = -0.21, 95% CI 2-sided [-4.85 to 4.43]
Statistical Analysis 2: Comparison: Boostrix + Menactra Group vs Menactra-Boostrix Group; Non-inferiority of Menactra™ vaccine co-administered with Boostrix® vaccine compared to Menactra™ vaccine administered alone at Month 0 with respect to a vaccine responseto meningococcal serogroup C one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was greater than the pre-defined limit of -10%; Difference in vaccine response rate = 1.69, 95% CI 2-sided [-1.69 to 5.16]
Statistical Analysis 3: Comparison: Boostrix + Menactra Group vs Menactra-Boostrix Group; Non-inferiority of Menactra™ vaccine co-administered with Boostrix® vaccine compared to Menactra™ vaccine administered alone at Month 0 with respect to a vaccine response to meningococcal serogroup Y one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was greater than the pre-defined limit of -10%; Difference in vaccine response rate = 1.82, 95% CI [-2.58 to 6.25]
Statistical Analysis 4: Comparison: Boostrix + Menactra Group vs Menactra-Boostrix Group; Non-inferiority of Menactra™ vaccine co-administered with Boostrix® vaccine compared to Menactra™ vaccine administered alone at Month 0 with respect to a vaccine response to meningococcal serogroup W-135 one month after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority objective was demonstrated if the lower limit was greater than the pre-defined limit of -10%; Difference in vaccine response rate = 3.56, 95% CI 2-sided [0.96 to 6.45]

5. Secondary Outcome: Number of Subjects With Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: Cut-off values assessed were greater than or equal to 1.0 international units per milliliter (IU/mL).
Time Frame: At Day 0 (PRE) before Boostrix vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 427 | 416 | 431
Participants
  ANTI-D, PRE: number analyzed (Participants) | 427 | 415 | 431
  ANTI-D, PRE | 109 | 93 | 120
  ANTI-T, PRE | 201 | 181 | 195

6. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: Cut-off values assessed were greater than or equal to 1.0 international units per milliliter (IU/mL).
Time Frame: At Month 2 (one month post Boostrix vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Menactra-Boostrix Group: Subjects, 11 through 18 years of age, received one dose of Menactra vaccine at Day 0 followed by one dose of Boostrix® vaccine at Month 1. Both vaccines were administered intramuscularly into the left deltoid region.
Arm/Group | Menactra-Boostrix Group
Number analyzed (Participants) | 429
Participants
  Anti-D | 428
  Anti-T | 426

7. Secondary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Antigens
Description: Cut-off values assessed were greater than or equal to 0.1 international units per milliliter (IU/m L).
Time Frame: PRE (Day 0) and POST Boostrix vaccination (Month 1 for Boostrix + Menactra Group and Boostrix-Menactra Group/ Month 2 for Menactra-Boostrix Group)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 428 | 416 | 431
Participants
  Anti-D, PRE: number analyzed (Participants) | 427 | 415 | 431
  Anti-D, PRE | 399 | 383 | 391
  Anti-T, PRE: number analyzed (Participants) | 427 | 416 | 431
  Anti-T, PRE | 423 | 409 | 423
  ANTI-D, POST: number analyzed (Participants) | 428 | 415 | 429
  ANTI-D, POST | 428 | 415 | 429
  ANTI-T, POST: number analyzed (Participants) | 428 | 415 | 429
  ANTI-T, POST | 428 | 415 | 429

8. Secondary Outcome: Number of Subjects With Booster Responses for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: Booster responses for anti-D and anti-T antibodies were defined as:
  for initially seronegative subjects (pre-vaccination concentration below the cut-off concentration of 0.1 IU/mL): antibody concentrations at least four times the cut-off (postvaccination concentration ≥ 0.4 IU/mL), one month after vaccination with the Boostrix vaccine; and for initially seropositive subjects (pre-vaccination concentration ≥ 0.1 IU/mL): an increase in antibody concentrations of at least four times the pre-vaccination concentration one month after vaccination with the Boostrix vaccine.
Time Frame: At one month POST Boostrix vaccination (Month 1 for Boostrix + Menactra Group and Boostrix-Menactra Group/ Month 2 for Menactra-Boostrix Group)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 427 | 414 | 428
Participants
  Anti-D, Total: number analyzed (Participants) | 427 | 413 | 428
  Anti-D, Total | 422 | 377 | 422
  Anti-T, Total | 310 | 330 | 329

9. Secondary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: PRE (Day 0) and one month POST Boostrix vaccination (Month 1 for Boostrix + Menactra Group and Boostrix-Menactra Group/ Month 2 for Menactra-Boostrix Group)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 428 | 416 | 431
IU/mL
  Anti-D, PRE: number analyzed (Participants) | 427 | 415 | 431
  Anti-D, PRE | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.5] | 0.5 [0.4 to 0.5]
  Anti-D, POST: number analyzed (Participants) | 428 | 415 | 429
  Anti-D, POST | 40.1 [36.9 to 43.5] | 10.2 [9.3 to 11.2] | 27.3 [25.1 to 29.6]
  Anti-T, PRE: number analyzed (Participants) | 427 | 416 | 431
  Anti-T, PRE | 1.0 [0.9 to 1.1] | 0.8 [0.8 to 0.9] | 0.9 [0.8 to 1.0]
  Anti-T, POST: number analyzed (Participants) | 428 | 415 | 429
  Anti-T, POST | 9.5 [8.9 to 10.2] | 12.7 [11.8 to 13.8] | 12.2 [11.3 to 13.2]

10. Secondary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: as for outcome 9
Time Frame: At one month POST Menactra vaccination (Month 2 for Boostrix-Menactra Group and Month 1 for Menactra-Boostrix Group)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 411 | 430
IU/mL
  Anti-D | 16.5 [15.4 to 17.6] | 41.6 [38.1 to 45.5]
  Anti-T | 10.0 [9.2 to 10.8] | 0.9 [0.8 to 1.0]

11. Secondary Outcome: Number of Subjects With Booster Responses for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies
Description: Booster responses for anti-PT, anti-FHA and anti-PRN antibodies were defined as: for initially seronegative subjects (pre-vaccination concentration below the cut-off concentration of 5 EL.U/mL): antibody concentrations at least four times the cut-off (postvaccination concentration ≥20 EL.U/mL) one month after vaccination with the Boostrix vaccine; for initially seropositive subjects with pre-vaccination concentration ≥5 EL.U/mL and < 20 EL.U/mL: an increase in antibody concentrations of at least four times the pre-vaccination concentration, one month after vaccination with the Boostrix vaccine; and for initially seropositive subjects with pre-vaccination concentration ≥ 20 EL.U/mL: an increase in antibody concentrations of at least two times the pre-vaccination concentration one month after vaccination with the Boostrix vaccine.
Time Frame: At Month 2 (one month post Boostrix vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra-Boostrix Group
Number analyzed (Participants) | 428
Participants
  Anti-PT, Total: number analyzed (Participants) | 423
  Anti-PT, Total | 338
  Anti-FHA, Total: number analyzed (Participants) | 424
  Anti-FHA, Total | 405
  Anti-PRN, Total | 414

12. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: At Day 0 before (PRE) Boostrix vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 427 | 416 | 431
EL.U/mL
  Anti-PT: number analyzed (Participants) | 419 | 412 | 428
  Anti-PT | 8.6 [7.7 to 9.6] | 10.0 [8.9 to 11.3] | 10.3 [9.2 to 11.6]
  Anti-FHA: number analyzed (Participants) | 425 | 414 | 428
  Anti-FHA | 46.5 [41.4 to 52.3] | 43.8 [39.1 to 49.0] | 47.8 [42.4 to 53.8]
  Anti-PRN | 12.5 [11.1 to 14.1] | 10.6 [9.3 to 12.0] | 12.0 [10.6 to 13.5]

13. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 2 (one month post Boostrix vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Menactra-Boostrix Group
Number analyzed (Participants) | 429
EL.U/mL
  Anti-PT: number analyzed (Participants) | 427
  Anti-PT | 77.8 [71.5 to 84.6]
  ANTI-FHA: number analyzed (Participants) | 428
  ANTI-FHA | 653.0 [603.6 to 706.5]
  Anti-PRN | 412.5 [364.5 to 466.9]

14. Secondary Outcome: Titers for rSBA-MenA, rSBA-MenC, rSBA-MenY and rSBA-MenW-135 Antibodies
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: PRE (Day 0) and one month POST Menactra vaccination (Month 2 for Boostrix + Menactra Group and Boostrix-Menactra Group / Month 1 for Menactra-Boostrix Group)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 424 | 408 | 427
Titers
  rSBA-MenA, PRE: number analyzed (Participants) | 379 | 357 | 381
  rSBA-MenA, PRE | 533.4 [464.6 to 612.3] | 490.8 [428.4 to 562.3] | 449.4 [383.4 to 526.6]
  rSBA-MenA, POST: number analyzed (Participants) | 421 | 394 | 420
  rSBA-MenA, POST | 10406.1 [9687.2 to 11178.3] | 7220.0 [6613.3 to 7882.4] | 9466.3 [8765.6 to 10222.9]
  rSBA-MenC, PRE: number analyzed (Participants) | 418 | 405 | 417
  rSBA-MenC, PRE | 21.0 [17.2 to 25.5] | 16.4 [13.6 to 19.8] | 18.7 [15.3 to 22.8]
  rSBA-MenC, POST: number analyzed (Participants) | 423 | 408 | 427
  rSBA-MenC, POST | 2760.2 [2387.5 to 3191.1] | 1137.0 [969.6 to 1333.3] | 2702.8 [2292.6 to 3186.5]
  rSBA-MenY, PRE: number analyzed (Participants) | 418 | 405 | 413
  rSBA-MenY, PRE | 53.8 [43.6 to 66.5] | 51.4 [41.6 to 63.5] | 56.2 [45.1 to 70.1]
  rSBA-MenY, POST: number analyzed (Participants) | 423 | 408 | 427
  rSBA-MenY, POST | 3244.2 [2884.1 to 3649.1] | 1470.7 [1311.4 to 1649.3] | 3022.8 [2687.0 to 3400.6]
  rSBA-MenW-135, PRE: number analyzed (Participants) | 416 | 395 | 422
  rSBA-MenW-135, PRE | 23.7 [19.5 to 28.6] | 28.0 [23.1 to 34.0] | 32.2 [26.6 to 39.0]
  rSBA-MenW-135, POST | 4822.1 [4351.6 to 5343.4] | 2143.1 [1913.9 to 2399.8] | 4154.3 [3690.9 to 4675.9]

15. Secondary Outcome: Number of Subjects With Vaccine Responses for rSBA-MenA, rSBA-MenC, rSBA-MenY and rSBA-MenW-135 Antibodies
Description: Vaccine responses for rSBA-MenA, rSBA-MenC, rSBA-MenY and rSBA-MenW-135 antibodies were defined as: for initially seronegative subjects (pre-vaccination concentration below the cut-off titer of 8): antibody titers at least four times the cut-off (post-vaccination concentration ≥ 32) one month after vaccination with Menactra the vaccine, and for initially seropositive subjects (pre-vaccination titer ≥ 8): antibody titers at least four times the pre-vaccination antibody titers, one month after vaccination with the Menactra vaccine.
Time Frame: At Month 2 (one month after vaccination with Menactra vaccine)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Menactra Group
Number analyzed (Participants) | 396
Participants
  rSBA-MenA, Total: number analyzed (Participants) | 339
  rSBA-MenA, Total | 300
  rSBA-MenC, Total | 351
  rSBA-MenY, Total | 325
  rSBA-MenW-135, Total: number analyzed (Participants) | 386
  rSBA-MenW-135, Total | 360

16. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = any solicited local symptom irrespective of intensity grade. Grade 3 pain = pain that prevented normal activities. Grade 3 redness/swelling = redness/swelling with diameter ≥ 50 millimeters (mm).
Time Frame: Within 4-days (Day 0-3) after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and with the symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 441 | 433 | 446
Participants
  Pain, Any, Dose 1: number analyzed (Participants) | 441 | 432 | 446
  Pain, Any, Dose 1 | 331 | 304 | 236
  Pain, Grade 3, Dose 1: number analyzed (Participants) | 441 | 432 | 446
  Pain, Grade 3, Dose 1 | 26 | 14 | 6
  Redness, Any, Dose 1: number analyzed (Participants) | 441 | 432 | 446
  Redness, Any, Dose 1 | 118 | 111 | 84
  Redness, ≥ 50 mm, Dose 1: number analyzed (Participants) | 441 | 432 | 446
  Redness, ≥ 50 mm, Dose 1 | 10 | 1 | 4
  Swelling, Any, Dose 1: number analyzed (Participants) | 441 | 432 | 446
  Swelling, Any, Dose 1 | 99 | 78 | 56
  Swelling, ≥ 50 mm, Dose 1: number analyzed (Participants) | 441 | 432 | 446
  Swelling, ≥ 50 mm, Dose 1 | 8 | 7 | 5
  Pain, Any, Dose 2: number analyzed (Participants) | 441 | 426 | 441
  Pain, Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 260 | 211
  Pain, Grade 3, Dose 2: number analyzed (Participants) | 441 | 426 | 441
  Pain, Grade 3, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 13 | 4
  Redness, Any, Dose 2: number analyzed (Participants) | 441 | 426 | 441
  Redness, Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 85 | 79
  Redness, ≥ 50 mm, Dose 2: number analyzed (Participants) | 441 | 426 | 441
  Redness, ≥ 50 mm, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 8 | 2
  Swelling, Any, Dose 2: number analyzed (Participants) | 441 | 426 | 441
  Swelling, Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 64 | 53
  Swelling, ≥ 50 mm, Dose 2: number analyzed (Participants) | 441 | 426 | 441
  Swelling, ≥ 50 mm, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 9 | 3
  Pain, Any, Across doses | 331 | 343 | 291
  Pain, Grade 3, Across doses | 26 | 26 | 9
  Redness, Any, Across doses | 118 | 141 | 119
  Redness, ≥ 50 mm, Across doses | 10 | 8 | 6
  Swelling, Any, Across doses | 99 | 105 | 84
  Swelling, ≥ 50 mm, Across doses | 8 | 13 | 8

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as oral temperature equal to or above 37.5 degrees Celsius (°C)], headache and gastrointestinal symptoms [gastro sympt]. Any = any solicited general symptom irrespective of intensity grade or relationship to vaccination. Grade 3 = symptoms that prevented normal activities. Grade 3 Fever = temperature higher than (>) 39° C. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Gastrointestinal symptoms included nausea, vomiting, diarrhea and/or abdominal pain.
Time Frame: Within 4-days (Days 0-3) after each dose and across doses
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 446 | 446 | 449
Participants
  Fatigue, Any, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Fatigue, Any, Dose 1 | 150 | 139 | 114
  Fatigue, Grade 3, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Fatigue, Grade 3, Dose 1 | 13 | 9 | 5
  Fatigue, Related, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Fatigue, Related, Dose 1 | 120 | 113 | 86
  Fever (orally), Any, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Fever (orally), Any, Dose 1 | 23 | 15 | 21
  Fever (orally), Grade 3, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Fever (orally), Grade 3, Dose 1 | 2 | 1 | 0
  Fever (orally), Related, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Fever (orally), Related, Dose 1 | 20 | 8 | 16
  Gastro sympt., Any, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Gastro sympt., Any, Dose 1 | 67 | 63 | 60
  Gastro sympt, Grade 3, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Gastro sympt, Grade 3, Dose 1 | 4 | 4 | 2
  Gastro sympt, Related, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Gastro sympt, Related, Dose 1 | 46 | 41 | 36
  Headache, Any, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Headache, Any, Dose 1 | 150 | 133 | 116
  Headache, Grade 3, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Headache, Grade 3, Dose 1 | 12 | 12 | 7
  Headache, Related, Dose 1: number analyzed (Participants) | 441 | 433 | 446
  Headache, Related, Dose 1 | 127 | 104 | 85
  Fatigue, Any, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Fatigue, Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 103 | 90
  Fatigue, Grade 3, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Fatigue, Grade 3, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 5 | 3
  Fatigue, Related, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Fatigue, Related, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 83 | 70
  Fever (orally), Any, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Fever (orally), Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 14 | 10
  Fever (orally), Grade 3, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Fever (orally), Grade 3, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 1 | 1
  Fever (orally), Related, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Fever (orally), Related, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 9 | 9
  Gastro sympt., Any, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Gastro sympt., Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 46 | 34
  Gastro sympt., Grade 3, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Gastro sympt., Grade 3, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 1 | 3
  Gastro sympt., Related, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Gastro sympt., Related, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 32 | 24
  Headache, Any, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Headache, Any, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 95 | 75
  Headache, Grade 3, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Headache, Grade 3, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 2 | 2
  Headache, Related, Dose 2: number analyzed (Participants) | 446 | 426 | 441
  Headache, Related, Dose 2 | NA — Not applicable, as both vaccines were administered at the same timepoint. | 72 | 56
  Fatigue, Any, Across: number analyzed (Participants) | 441 | 434 | 446
  Fatigue, Any, Across | 150 | 175 | 160
  Fatigue, Grade 3, Across: number analyzed (Participants) | 441 | 434 | 446
  Fatigue, Grade 3, Across | 13 | 13 | 7
  Fatigue, Related, Across: number analyzed (Participants) | 441 | 434 | 446
  Fatigue, Related, Across | 120 | 146 | 128
  Fever (orally), Any, Across: number analyzed (Participants) | 441 | 434 | 446
  Fever (orally), Any, Across | 23 | 28 | 29
  Fever (orally), Grade 3, Across: number analyzed (Participants) | 441 | 434 | 446
  Fever (orally), Grade 3, Across | 2 | 2 | 1
  Fever (orally), Related, Across: number analyzed (Participants) | 441 | 434 | 446
  Fever (orally), Related, Across | 20 | 16 | 23
  Gastro sympt., Any, Across: number analyzed (Participants) | 441 | 434 | 446
  Gastro sympt., Any, Across | 67 | 96 | 80
  Gastro sympt., Grade 3, Across: number analyzed (Participants) | 441 | 434 | 446
  Gastro sympt., Grade 3, Across | 4 | 5 | 5
  Gastro sympt., Related, Across: number analyzed (Participants) | 441 | 434 | 446
  Gastro sympt., Related, Across | 46 | 65 | 54
  Headache, Any, Across: number analyzed (Participants) | 441 | 434 | 446
  Headache, Any, Across | 150 | 177 | 157
  Headache, Grade 3, Across: number analyzed (Participants) | 411 | 434 | 446
  Headache, Grade 3, Across | 12 | 13 | 9
  Headache, Related, Across: number analyzed (Participants) | 441 | 434 | 446
  Headache, Related, Across | 127 | 142 | 121

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE =An AE which prevented normal, everyday activities. Such an AE, for example, prevented attendance at work/school and necessitated the administration of corrective therapy. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 31-day (Days 0-30) period after each vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 446 | 446 | 449
Participants
  Any AEs | 124 | 149 | 155
  Grade 3 AEs | 16 | 15 | 22
  Related AEs | 37 | 44 | 29

19. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the entire study period (Day 0 - Month 2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Number analyzed (Participants) | 446 | 446 | 449
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms during the 4-day (Day 0-3) follow-up period, unsolicited AEs during the 31-day (Day 0-30) follow-up period after each vaccination and SAEs throughout the study (Day 0 - Month 2).
Groups:
- Boostrix + Menactra Group: Subjects, 11 through 18 years of age, received a booster dose of Boostrix® co-admisistered with Menactra™ at Day 0. The Boostrix® vaccine was administered intramuscularly into the left deltoid region and Menactra™ vaccine was administered intramuscularly into the right deltoid region.
Arm/Group | Boostrix + Menactra Group | Boostrix-Menactra Group | Menactra-Boostrix Group
Serious Adverse Events (participants affected / at risk) | 1/446 | 0/446 | 1/449
Other Adverse Events (participants affected / at risk) | 371/446 | 385/446 | 358/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix + Menactra Group (N=446) | Boostrix-Menactra Group (N=446) | Menactra-Boostrix Group (N=449)
Extradural hematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix + Menactra Group (N=446) | Boostrix-Menactra Group (N=446) | Menactra-Boostrix Group (N=449)
Pain (General disorders) | 331 | 343 | 291
Redness (General disorders) | 118 | 141 | 119
Swelling (General disorders) | 99 | 105 | 84
Fatigue (General disorders) | 150 | 175 | 160
Fever (orally) (General disorders) | 23 | 28 | 29
Gastrointestinal symptoms (General disorders) | 67 | 96 | 80
Headache (General disorders) | 150 | 177 | 157

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.